CLINICAL TRIAL: NCT06523452
Title: The Clinical and Cost Effectiveness of Intra-operative Laser Speckle Imaging (LSI) of Tissue Blood Flow to Avoid Post-operative Complications Following Breast Reconstruction After Mastectomy for Breast Cancer: A Feasibility Study
Brief Title: Laser Speckle Imaging During Breast Reconstruction
Acronym: SIMBAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2405577
Record Dates: First submitted 2024-06-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSI Assisted Group (Experimental): Breast reconstruction surgery will be standard clinical care, but tissue blood flow images will be available during surgery to aid surgical decision making.
  The surgical procedure will take slightly longer (approximately 10-15 minutes in total) compared to the Treatment As Usual group.
  Interventions: Other: Laser Speckle Imaging
- Treatment As Usual Group (No Intervention): Breast reconstruction surgery will be standard clinical care

INTERVENTIONS:
Other: Laser Speckle Imaging — At least three scans (four for skin sparing mastectomy) will be performed on participants randomised to the LSI Assisted Group. Further scans may be taken at the discretion of the surgeon.
  Arms: LSI Assisted Group

SUMMARY:
Around 3500 women a year have surgery to reconstruct a breast/s after cancer. Breast reconstruction can have a positive impact on their lives, but unfortunately 3 or 4 in 10 women have problems with healing after their operation. This is distressing and often leads to more medical care or surgery. These problems are often caused by poor blood flow to the skin and deeper tissues used to reconstruct the breast. The investigators have developed a new device that does not touch the skin and provides immediate, continuous images of skin blood flow (the flow that surgeons cannot see). To test this device the investigators took images of blood flow during breast reconstruction surgery. The investigators found that imaging was good at showing where skin blood flow was poor and led to problems with healing and where flow was good and there were fewer problems after surgery (from minor problems, e.g. delayed healing; to major problems, e.g. loss of new breast).

The investigators think this device can help surgeons choose healthy skin during breast reconstruction and so help more patients to heal without surgical problems. The investigators need to test the new imaging device in a large clinical trial to find out how effective it is at improving healing for women after breast reconstruction. Before this, the investigators need to find out if such a trial is possible and acceptable to patients, theatre staff and surgeons. The investigators will recruit 60 women who are having breast surgery and will randomly choose 30 to have surgery without blood flow imaging and 30 to have surgery with blood flow imaging. The investigators will follow up the women whilst in hospital and for the following 6 months to record any problems. In particular the investigators need to find out how many patients will volunteer for the study and the study can collect all the information needed during the 6 months after surgery. The results from this study will be used to plan a much larger clinical trial that will test whether blood flow imaging is effective, improves patient recovery after surgery and provides good value for money for the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 or over;
* Able and willing to provide informed consent;
* Scheduled for breast reconstruction by autologous free flap surgery (either immediately post-mastectomy or delayed).

Exclusion Criteria:

* Unable to give written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rate for both LSI-Assisted and TAU groups | End of Trial - 6 months after entry of final participant
  Number of participants recruited to the study and number lost to follow up
Rates of post-operative complications for both LSI and TAU groups | End of Trial - 6 months after entry of final participant
  Number of participants with post-operative complications and their severity over 6 months post operative using patient diaries and patient notes assessed by Clavien-Dindo or CTCAE.

SECONDARY OUTCOMES:
A health economic framework for the future trial. | End of Trial - 6 months after entry of final participant
  Economic evaluation methods will be developed and tested on the collection of resource use, cost and QoL outcome data assessed using Resource Use, EQ-5D-5L and BREAST Q questionnaires.
LSI training manual and understanding the views of theatre staff on the use of LSI. | End of Trial - 6 months after entry of final participant
  Develop appropriate training material for use of LSI Device through conducting pre-operative observations, focus groups and post operative interviews with theatre staff to assess feasibility and acceptability of LSI.
Understanding the views of patients on the use of LSI. | End of Trial - 6 months after entry of final participant
  Conduct qualitative interviews with patients in both LSI and TAU groups
LSI perfusion measures in the two groups | End of Trial - 6 months after entry of final participant
  Assess the perfusion through the

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No